CLINICAL TRIAL: NCT01163682
Title: Randomized Sham Controlled Trial of Weekly Electro-acupuncture for the Prevention of Taxane Induced Myalgias and Neuropathy
Brief Title: Electro-acupuncture for the Prevention of Taxane Induced Myalgias and Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Dawn L. Hershman, Associate Professor of Medicine & Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AAAE7054
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; Neuropathy
Keywords: taxane induced neuropathy; taxane induced myalgias; electro-acupuncture
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Electro-acupuncture (Experimental): Subjects will receive 45 minute sessions scheduled once a week for 12 weeks with electro-acupuncture.
  Interventions: Device: Electro-acupuncture
- Sham acupuncture (Sham Comparator): Subjects will receive 45 minute sessions scheduled once a week for 12 weeks with sham acupuncture.
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Electro-acupuncture — Subjects will be placed in prone position and acupuncture sites will be cleaned with alcohol preparation. Stainless steel disposable acupuncture needle (diameter 0.25mm) will be inserted into the skin to appropriate depth needed to elicit de qi(approximately 3-4mm). Selected acupuncture points will be attached to2 leads connected to an electro-stimulator that generates 2 Hz of mixed pulsatile intervals for a total of 30 minutes. The acupuncturist will return two times during the treatment at 10 and 20 minutes with needles in situ to check on the patients and needles. Needles not attached to the electro-stimulator will be manipulated manually to elicit de qi one time during the treatment.
  Arms: Electro-acupuncture
Device: Sham acupuncture — Will be utilizing a sham control that consists of collapsible acupuncture needle so that there is no penetration of skin. The sham needles will be place on 4 non specific body points. The electro-stimulator will be attached to the needles for 30 minutes but will not be turned on. The acupuncturist will return two times during the treatment at 10 and 20 minutes to check on the patient. The acupuncturist will touch the collapsible acupuncture needs to simulate the manipulation of the needles.
  Arms: Sham acupuncture

SUMMARY:
This study seeks to determine if 12 weeks of weekly electro-acupuncture will prevent or decrease neuropathic pain in breast cancer patients receiving 12 weekly treatments of taxane treatment.

DETAILED DESCRIPTION:
Chemotherapy induced neuropathy (CIN) is a common and disabling toxicity of cytotoxic chemotherapy. Depending on the drug, it is often irreversible even after the offending agent is removed. The consequence of terminating effective anti-tumor therapy or dose reduction can be catastrophic to the effect of a patient's cancer treatment. Given the morbidity of taxane induced neuropathy, the lack of effective preventative treatment for taxane induce neuropathy and the safety of acupuncture, it is reasonable to test the efficacy of this non pharmacological intervention in woman with Stage I-III breast cancer receiving adjuvant or neo-adjuvant weekly paclitaxel for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age>21 years
* History of stage I-III breast cancer
* Patient scheduled to be receiving weekly adjuvant or neo-adjuvant paclitaxel for 12 weeks
* Signed informed consent

Exclusion Criteria:

* Previous treatment with acupuncture in the last 12 months
* Diabetic Neuropathy or other neurological conditions
* Inflammatory, metabolic or neuropathic arthropathies
* Current narcotic use
* Severe concomitant illnesses
* Severe coagulopathy or bleeding disorder
* Dermatological disease within the acupuncture area
* Have a pacemaker

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn L Hershman, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 180 participants were screened, of which 99 refused to take part in the study, 16 were ineligible, and 2 withdrew before the intervention began. 63 participants were enrolled and randomized to the two treatment groups.
Period: Overall Study
Arm/Group | Electro-acupuncture | Sham Acupuncture
Started | 31 | 32
Completed | 25 | 23
Not Completed | 6 | 9
Not completed — Lost to Follow-up | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electro-acupuncture | Sham Acupuncture | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.8 (10.7) | 48.3 (12.0) | 50.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 13 | 14 | 27
  Non-hispanic White | 7 | 9 | 16
  African America | 10 | 6 | 16
  Asian | 1 | 3 | 4
Breast Cancer Type [Count of Participants; unit: Participants]
  Invasive ductal carcinoma | 25 | 27 | 52
  Invasive lobular carcinoma | 5 | 5 | 10
  Sarcomatoid | 1 | 0 | 1
ER/PR status [Count of Participants; unit: Participants]
  Negative | 7 | 8 | 15
  Positive | 24 | 24 | 48
HER2 status [Count of Participants; unit: Participants]
  Negative | 25 | 22 | 47
  Positive | 6 | 10 | 16
Breast Cancer Stage [Count of Participants; unit: Participants] — Breast cancer staging performed based on standard of care diagnostic procedures outside of this trial. A lower breast cancer stage (Stage 1) indicates a less advanced stage of cancer.
  Participants
    Stage I Breast Cancer | 2 | 4 | 6
    Stage II Breast Cancer | 26 | 19 | 45
    Stage III Breast Cancer | 3 | 9 | 12
Tumor Grade [Count of Participants; unit: Participants]
  Well differentiated | 2 | 0 | 2
  Moderately differentiated | 14 | 15 | 29
  Poorly differentiated | 15 | 17 | 32
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (6.3) | 29.5 (7.1) | 28.6 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Brief Pain Inventory-Short Form Score
Description: The change in neuropathic pain, as measured by the mean Brief Pain Inventory-Short Form (BPI-SF) worst pain score, from baseline to 16 weeks, in the study group that received electro-acupuncture (intervention), was compared to the change in neuropathic pain in the study group that received sham acupuncture (control). Scores range from 0 (no pain)-10 (worst pain) with a higher score indicating worse outcome.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Electro-acupuncture | Sham Acupuncture
Number analyzed (Participants) | 25 | 23
Score on a scale | 1.6 (3) | 0.6 (2.1)
Statistical Analysis 1: Comparison: Electro-acupuncture vs Sham Acupuncture; Test type: Non-Inferiority — This tests determined the odds of an increase of greater than or equal to 2 points on the BPI-SF worst pain score, from baseline to 16 weeks, among those in the intervention arm (electo-acupuncture), compared to those in the control arm (sham acupuncture). This change was considered to be clinically meaningful. Null Hypothesis: electro-acupucture does not prevent taxane-induced peripheral neuropathy; p = 0.25, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.90 to 1.50]

2. Secondary Outcome: Change in FACT-TAX Score
Description: The change in the quality of life as measured by Functional Assessment of Cancer Therapy- Taxane (FACT-TAX) quality of life assessment, collected at baseline and 16 weeks, as compared between the intervention and control study groups (electro acupuncture and sham acupuncture). is a validated self reported instrument used to measure self reported neuropathic symptoms among patients undergoing taxane therapy. There are four quality of life (QOL) domains as part of the FACT that include physical well being, social well being, emotional well being and functional well being. The taxane subscale combines a validated 11 item neurotoxicity subscale with 5 additional questions assessing symptoms related to arthralgias, myalgias and skin changes. The FACT-TAX scale ranges from 0-64 with five response levels (0= very much, 4 = not at all). Higher scores indicate better quality of life or fewer symptoms.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Electro-acupuncture | Sham Acupuncture
Number analyzed (Participants) | 25 | 23
Score on a scale | -9.4 (11) | -8.4 (9.8)
Statistical Analysis 1: Comparison: Electro-acupuncture vs Sham Acupuncture; Test type: Non-Inferiority — This tests determined the odds of an increase of greater than or equal to 5 points on the FACT-NTX scale, from baseline to 16 weeks, among those in the intervention arm (electo-acupuncture), compared to those in the control arm (sham acupuncture). This change was considered to be clinically meaningful; p = 0.09, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.97 to 1.62]

ADVERSE EVENTS:
Arm/Group | Electro-acupuncture | Sham Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 1/31 | 0/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electro-acupuncture (N=31) | Sham Acupuncture (N=32)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0) — A grade 1 acupuncture needle site reaction with discomfort, minor swelling, and bruising after acupuncture needle withdrawal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes